CLINICAL TRIAL: NCT03076294
Title: Repetitive Transcranial Magnetic Stimulation Associated With Manual Therapy in Knee Ostearthritis Pain
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Universidade Federal de Pernambuco (Other)
Responsible Party: Principal Investigator, Kátia Monte-Silva, PhD, Universidade Federal de Pernambuco
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: OA_TMS_Pain
Record Dates: First submitted 2017-03-06; First posted 2017-03-10 (Actual); Last update posted 2017-03-10 (Actual); Status verified 2017-03

CONDITIONS: Knee Osteoarthritis
Keywords: knee ostearthritis; transcranial magnetic stimulation; repetitive transcranial magnetic stimulation; chronic pain; musculoskeletal manipulations
MeSH Terms: conditions — Osteoarthritis, Knee; Chronic Pain | interventions — Musculoskeletal Manipulations

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- MT after rTMS group (Experimental): High frequency TMS will be applied with an eight-shaped coil angled at zero degrees from the sagittal axis and positioned at the C3 or C4 in accordance with the international 10-20 marking system (JASPER, 1958), which corresponds to the right or left primary motor cortex (M1). Twenty four stimulus trains will be provided at 10 Hz for five seconds each. The interval between the trains will be 25 seconds, totaling 1200 pulses for approximately 12 minutes, with 90% of resting motor threshold (RMT). After TMS, patients will be submitted to 45 minutes of manual therapy protocol.
  Interventions: Device: TMS; Other: Manual therapy (MT)
- rTMS after MT group (Experimental): Patients will be submitted to 45 minutes of manual therapy protocol. After that, high frequency TMS will be applied with an eight-shaped coil angled at zero degrees from the sagittal axis and positioned at the C3 or C4 in accordance with the international 10-20 marking system (JASPER, 1958), which corresponds to the right or left primary motor cortex (M1). Twenty four stimulus trains will be provided at 10 Hz for five seconds each. The interval between the trains will be 25 seconds, totaling 1200 pulses for approximately 12 minutes, with 90% of resting motor threshold (RMT).
  Interventions: Device: TMS; Other: Manual therapy (MT)
- Control group (Sham Comparator): In this group, the order of interventions will be randomized. Therefore, the volunteer can start with manual therapy or sham TMS. In manual therapy, patients will be submitted to 45 minutes of a protocol. In addition, with regard to sham TMS, the same parameters will be used, however, it will be performed using two coils, one connected to the magnetic stimulator, away from the patient's scalp and another uncoupled from the stimulator and positioned in the same way as in real stimulation.
  Interventions: Device: TMS; Other: Manual therapy (MT)

INTERVENTIONS:
Device: TMS — Repetitive TMS involves application of electric currents in the patient's cortex by a magnetic field applied to the scalp of the patient through an eight-coil connected to a magnetic stimulator (MagStim Rapid² magnetic stimulator-UK). In a small percentage of patients, it may cause minimal discomfort with a mild headache sensation, which usually disappears after a few seconds. Depending on the parameters, rTMS can increase or decrease corticomotor excitability and by the connection of the motor cortex with the thalamus, influencing pain control. The patients will respond to an adverse effects questionnaire and will report the perception of real or sham stimulation.
  Other Names: non invasive brain stimulation, high frequency TMS
Other: Manual therapy (MT) — This intervention uses manual contact for diagnosis and treatment, its practitioners use an enormous amount of manual techniques to preserve the homeostasis through the recovery of dysfunctions, which may cause limitations in the physiological movements, in the accessory movements of the joints (WHO , 2010).
  Other Names: Musculoskeletal manipulation

SUMMARY:
In this study, the investigators wondered whether the association between high frequency repetitive transcranial magnetic stimulation (hf-rTMS) and manual therapy (peripheral and central approach) is more effective in reducing pain levels and modulation of cortical activity of chronic knee ostearthritis pain subjects than manual therapy alone (usual peripheral approach). For this purpose, patients included will be submitted to one session with active or sham hf-rTMS followed by a protocol of manual therapy. Besides that another active group will have the sequence of interventions exchanged (manual therapy followed by hf-rTMS) in order to investigate whether this may influence in the final outcomes.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of knee OA;
* Absence of severe cognitive deficiency verified by the Mini Mental State Examination;
* Meet the American College of Rheumatology criteria for idiopathic knee osteoarthritis.

Exclusion Criteria:

* Individuals diagnosed with osteoporosis, fibromyalgia or other neurological disease;
* Had an opioid or corticosteroid injection in the last 30 days;
* Modified chronic pain medication in the last month before participating in the study;
* History of knee surgery in the last six months;
* Obese;
* Contraindications to the use of non-invasive brain stimulation, such as: metal implant on face or skull, history of seizure, cochlear implant.

Ages: 50 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 15 (Estimated)
Dates: Start 2017-01; Primary Completion 2018-03 (Estimated); Study Completion 2019-03 (Estimated)

PRIMARY OUTCOMES:
Pain | Until one day (before and after the interventions)
  Pain will be evaluated by pressure algometry before and after the interventions. It's a evaluation technique which aims to quantify through physical stimulation (pressure in the nociceptors) the capacity of pain perception and toleration. It will be used with the patient lying in supine and will have the purpose of measure the pressure pain threshold (PPT) in eight points around patellar region. Besides that, two control points will be adopted, one in anterior tibial muscle (five centimeters distal of anterior tibial tuberosity) and another in the extensor carpi radialis longus muscle (five centimeters distal to lateral humerus epicondyle). After marking, the algometer will be setted up 90° in contact with the skin and will be applied a 0,3 kgf/cm²/s pressure until the patient report pain by pressing a pen (Model/Brand: Algomed/Medoc). The measure will be done twice in the demarcated points with a two minutes interval between them. Will be considered a mean of the obtained values.
Pain Rating Scale (NPRS) | Until 30 days (before, after the interventions and until the last day with the same value of the first evaluation)
  Is it used to quantify pain level, where 0 means no pain and 10 means worst pain possible. NPRS is recommended as the main endpoint in chronic pain studies and it has been established that a decrease of at least 2 points or 30% represents a minimal clinically important difference. The MDCI consists of the smaller variation in a clinical outcome perceived by the patient and that results in a relevant change in his state of health.

SECONDARY OUTCOMES:
Cortical excitability | One day (before and after the interventions)
  The motor evoked potential (MEP) will be provided by twenty unconditioned stimuli (120% of motor resting threshould).

CONTACTS AND LOCATIONS:
Overall Officials: Kátia Monte-Silva, PhD, Study Director — Applied Neuroscience Laboratory, Universidade Federal de Pernambuco
Locations (2):
- Brazil (2):
  - Applied Neuroscience Laboratory, Universidade Federal de Pernambuco, Recife, Pernambuco
  - Kinesiotherapy and manual therapeutic resources laboratory, Recife, Pernambuco